CLINICAL TRIAL: NCT02437149
Title: Effectiveness of Distracted Driving Campaign for Teenagers in the Emergency Department
Brief Title: Effectiveness of Distracted Driving Campaign
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nicklaus Children's Hospital f/k/a Miami Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20150548
Record Dates: First submitted 2015-04-23; First posted 2015-05-07 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Trauma Prevention
Keywords: Texting and driving; Teenager and driving; Distracted Driving Campaign
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Video and Brochure (Experimental): Real stories video presentation and a brochure with information about distracted driving will be given to the participant.
  Interventions: Behavioral: Video; Behavioral: Brochure
- Power Point and Brochure (Experimental): Brief power point presentation and a brochure with information about distracted driving will be given to the participant.
  Interventions: Behavioral: Power Point; Behavioral: Brochure
- Brochure Only (Experimental): Only a brochure with information about distracting driving will be given to the participant.
  Interventions: Behavioral: Brochure

INTERVENTIONS:
Behavioral: Video — Real stories video presentation about distracted driving. Produced by the National Highway Traffic Safety Administration.
  Arms: Video and Brochure
Behavioral: Power Point — Brief power point presentation with information about distracted driving. Produced by the National Highway Traffic Safety Administration.
  Arms: Power Point and Brochure
Behavioral: Brochure — Brochure with the National Highway Traffic Safety Administration information about distracting driving.

SUMMARY:
The study will measure the effectiveness of a distracted driving campaign in the emergency department in teenagers, 15 to 18 years old, to determine if it changes their attitudes towards texting while driving. It will also assess previous knowledge and behaviors in this age group, regarding distracted driving and what educational tool (power point vs. videos vs. brochure) has the most impact changing the attitudes towards texting and driving.

DETAILED DESCRIPTION:
Distracted driving is defined by the National Highway Safety Administration (NHTSA) as any activity that could withdraw a person's attention away from the primary task of driving. It includes, talking or texting on a cell phone, grooming, eating or drinking, changing radio stations, or talking to passengers. Of all these activities text messaging is by far the most alarming distraction because it requires visual, manual, and cognitive attention from the driver.

The NHTSA Research Note on distracted driving found that in 2011, 10% percent of fatal crashes were reported as distraction-affected crashes. This research also showed that teens between 15 to 19 years old are currently the largest group with distracted driving affected crashes, with 21% percent of them getting distracted while using their cell phones.

During the last few years, multiple public awareness campaigns have been launched in attempt to reduce this problem. These massive campaigns have included television, radio and internet campaigns, posters, billboards and brochures among others. Nevertheless, there are no studies assessing the success of these methods.

The research project will use visual and verbal educational tools to engage this population in order to maximize the learning process. The project will include brochures, video presentations and power point presentations. The investigators intend to test a potentially new and effective way to teach our teenagers about the dangers of distracted driving. The project primary goal is to assess if a distracting driving campaign in the emergency department is effective in changing the attitudes towards texting while driving. The investigator also intends to assess the current knowledge about distracted driving and to determine which tool (visual vs. verbal) is most effective to deliver this message.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents between the ages of 15 to 18 years

Exclusion Criteria:

* Adolescents refusing to participate in the Distracted Driving Campaign.
* Adolescents visiting the emergency department with a chief complaint related to mental illness, suicide ideation or attempt, or any complaint limiting the ability to complete the questionnaire.
* Adolescents with diagnosis of developmental delay that could affect his or her ability to complete the questionnaire.
* Adolescents that do not speak English (the videos about real people who have had accidents while texting and driving found at http://www.distraction.gov/faces/index.html are available only in English.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 273 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Previous knowledge and attitudes towards distracted driving | 6 months
  A "Pre Campaign Survey" will be given to every participant before the intervention. The survey is a validated questionnaire that assess previous knowledge and attitudes towards distracted driving and demographic variables.

SECONDARY OUTCOMES:
Short Term Effectiveness of the Distracted Driving Campaign | 6 months
  A validated post campaign survey will be given, to each participant, immediately after the intervention. The "Post Campaign Survey 1" will assess the short term effectiveness of the campaign.
Long Term Effectiveness of the Distracted Driving Campaign | 6 months
  A "Post Campaign Survey 2" will be obtain by phone call, at least one month after the intervention is done, to assess long term effectiveness of the campaign.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Blumstein, MD, Principal Investigator — Nicklaus Children's Hospital f/k/a Miami Children's Hospital
Locations (1):
- Nicklaus Children's Hospital f/k/a Miami Children's Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided